CLINICAL TRIAL: NCT05780151
Title: Pan-European Proof-of-concept Study Comparing Decentralised Clinical Trial (DCT) and Hybrid Approaches to Conventional Clinical Trial Approaches in Patients With Type 2 Diabetes Mellitus Treated With Toujeo®
Brief Title: Remote And Decentralised Innovative Approaches to Clinical Trials (RADIAL)
Acronym: RADIAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mira Zuidgeest (Other)
Collaborators: IMI Trials@Home consortium (Unknown); Innovative Medicines Initiative (Other); Sanofi (Industry)
Responsible Party: Sponsor-Investigator, Mira Zuidgeest, Associate Professor, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EU-CT number 2022-500449-26-00; 1006010 (Other: Central Ethics Committee UK)
Record Dates: First submitted 2023-03-08; First posted 2023-03-22 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: decentralised clinical trial approach; proof-of-concept study
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Intervention Model Description: Parallel-group, open-label, multi-centre study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional (Active Comparator): In RADIAL, the main study intervention is a methodological intervention with patients being recruited into three arms with different level of decentralization. Additionally, participants in all arms are switching from their previously used basal insulin to Toujeo®, which is the clinical intervention, in the protocol defined as the study drug.
  The conventional arm is modelled after a previous clinical trial with a similar indication and intervention and aims to represent current state-of-the art clinical trial conduct.
  Interventions: Other: Methodological intervention; Drug: Toujeo
- Hybrid (Active Comparator): In RADIAL, the main study intervention is a methodological intervention with patients being recruited into three arms with different level of decentralization. Additionally, participants in all arms are switching from their previously used basal insulin to Toujeo®, which is the clinical intervention, in the protocol defined as the study drug.
  The hybrid trial design is defined as a trial containing conventional trial elements, such as site-based recruitment and screening visits, as well as decentralised trials elements, such as a remote follow-up period and data collection
  Interventions: Other: Methodological intervention; Drug: Toujeo
- Remote (Active Comparator): In RADIAL, the main study intervention is a methodological intervention with patients being recruited into three arms with different level of decentralization. Additionally, participants in all arms are switching from their previously used basal insulin to Toujeo®, which is the clinical intervention, in the protocol defined as the study drug.
  The remote arm is fully decentralised and aims to represent future decentralised clinical trial practice using a decentralised recruitment model, intervention period and data collection.
  Interventions: Other: Methodological intervention; Drug: Toujeo

INTERVENTIONS:
Other: Methodological intervention — All three arms will receive the same clinical intervention but will differ in their level of decentralisation, the methodological intervention.
Drug: Toujeo — All participants in the study will receive Toujeo® (insulin glargine 300 U/mL). During the treatment period, Toujeo® injection will be administered once daily at the same time as the participant's previous basal insulin was injected, for participant previously treated with once daily injection. In case of previous insulin treatment administered twice a day, the time of injection of Toujeo® will have to be agreed between the physician and the participant before first administration.
  Other Names: insulin glargine 300 U/ml

SUMMARY:
Pan-European proof-of-concept study comparing Decentralised Clinical Trial (DCT) and hybrid approaches to conventional clinical trial approaches in patients with Type 2 diabetes mellitus treated with Toujeo®.

DETAILED DESCRIPTION:
The proposed study has been designed to compare the scientific and operational quality of fully decentralised and hybrid approaches to a conventional clinical trial approach and evaluate the feasibility of such approaches.

The primary study objectives are to (1) assess potential benefits of a DCT approach on participant recruitment, retention, diversity, site and participant satisfaction, and cost and (2) to determine acceptability of a DCT approach by measuring variables related to safety oversight, treatment adherence and data quality (missing data and query rate) within the arms that have a different degree of decentralisation.

The secondary study objective is to determine whether the efficacy of treatment with Toujeo® (insulin glargine 300 U/mL) is within the accepted range within the arms with different degree of decentralisation.

The design is a parallel-group, open-label, multi-centre study in Europe for patients with Type 2 diabetes mellitus ( T2DM) with glycated haemoglobin (HbA1c) between 7% and 10% and treated with basal insulin as part of their glucose-lowering treatment. The study consists of 2 parts with 3 different arms. Part A has site-based recruitment followed by a 1:1 randomization into a conventional arm and a hybrid arm. Part B has decentralised recruitment, no randomization and consists of a fully remote arm.

The study will enrol approximately 150 adults in each site-based arm (conventional and hybrid) and approximately 300 in the remote arm, for a total of 600 participants in approximately 5-6 countries. Both Part A and Part B will consist of a screening period (3-6 weeks), a treatment period with open-label Toujeo® (24 weeks) and a follow-up period (2-4 days after end of treatment [EOT]).

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

1. Participant with T2DM diagnosed for at least 1 year before the screening visit (V1).
2. Participant treated with a stable basal insulin regimen (i.e. type of insulin and time/frequency of the injection), for at least 3 months before the screening visit.
3. The total daily basal insulin dose should be stable (±20%) for at least 1 month before the screening visit.
4. Participant treated with ≥1 noninsulin antidiabetic drugs at stable dose in the 3 months before the screening visit.
5. Signed written informed consent or e-consent depending on the arm.
6. Participant's mental and physical status allows them to be able to perform their activities of daily living with no or minimal assistance, including the ability to administer injectable insulin and measure their blood glycaemic level.
7. Willing and able to permit home visits (only for Part A of the study).
8. Willing and able to comply with study drug receipt, accountability, and return processes and procedures.
9. Access to tablet/smartphone with Bluetooth functionality.
10. Access to internet connection that allows remote data entry and, for part B, video conferencing.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

1. Age <18 years.
2. HbA1c at screening visit: <7.0% or >10.0%.
3. Patient not willing to self-manage insulin titration algorithm.
4. Type 1 diabetes mellitus.
5. Treatment with mixed insulin (premixes), short-acting insulin, fast acting insulin analogues or Toujeo® during the 3 months before the screening visit.
6. Use of systemic glucocorticoids (excluding topical application or inhaled forms) for two weeks or more within 8 weeks prior to the time of screening.
7. Any clinically significant abnormality identified at the time of screening, or any condition (including known substance or alcohol abuse, or psychiatric disorder) that in the opinion of the Investigator or any sub-Investigator would make implementation of the protocol or interpretation of the study results difficult or would preclude the safe participation of the participant in this study.
8. Use of any investigational drug within 1 month or 5 half-lives, whichever is longer, prior to screening visit.
9. Participant is the Investigator or any Subinvestigator, research assistant, pharmacist, study coordinator, other staff or relative thereof directly involved in the conduct of the protocol.
10. Participant whom the investigator deems otherwise ineligible (e.g. unable to understand and follow instructions). Reason for ineligibility will be documented.
11. Pregnant or breastfeeding woman at the time of screening.
12. Woman of childbearing potential not protected by acceptable method(s) of birth control and/or who are unwilling or unable to be tested for pregnancy (see Section 10.3).
13. Known hypersensitivity / intolerance to insulin glargine or any of Toujeo® excipients.
14. Participant who withdraws consent during the screening (participant who is not willing to continue or fails to return).
15. Despite screening of the participant, enrolment is stopped at the study level.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2025-01-21 (Actual); Study Completion 2025-01-21 (Actual)

PRIMARY OUTCOMES:
Enrolment rates | 32 weeks
  Time to enrolment from Site activation until last participant enrolled
Retention rates | 6 months
  Proportion of participants completing the study period
Diversity | 10 weeks
  Various diversity aspects such as race, ethnicity, socioeconomic status, digital literacy, distance to health care professional, mobility.
Participant satisfaction | 6 months
  Participant satisfaction measured using a questionnaire just after V2 (baseline), V6 and V9 (EOT)
Site staff satisfaction | 6 months
  Site staff satisfaction measured using a questionnaire (after study initiation visit [SIV]), after 3 enrolled participants, after 3 participants completed Week 12 and after last patient last visit (LPLV).
Study cost | complete trial duration
  Absolute cost per participant using a combination of prospective and retrospective measurements
Time of AE (Adverse Event)/ SAE (Serious Adverse Event) occurence to collection | 6 months
  Time from event occurrence to collection AE/SAE in the eDiary or eCRF (electronic Case Report Form), whichever is applicable.
Treatment adherence | 6 months
  Adherence to the daily insulin injection by means of eDiary analysis in percentage of days of documented intake until participant's EOT.
Missing data | 9 months
  Proportion of missing data on the critical data points (Hb1Ac, Fasting Glucose, Participant satisfaction questionnaire)
Query rate | 9 months
  Number of queries (both manual and automatic) per participant per arm.

CONTACTS AND LOCATIONS:
Overall Officials: Mira GP Zuidgeest, PhD, Principal Investigator — UMC Utrecht
Locations (9):
- Denmark (2):
  - Steno Diabetes Centre Odense, Odense
  - Syddansk Universitet, Odense
- Germany (3):
  - Studienzentrum Diabetespraxis Dr. Braun, Berlin
  - Klinische Forschung Dresden GmbH, Dresden
  - Velocity Clinical Research Leipzig GmbH, Leipzig
- United Kingdom (4):
  - FutureMeds Soho Health Centre, Birmingham
  - Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool
  - University Hospitals Leicester NHS Trust, Leicester
  - NIHR Patient Recruitment Centre Newcastle, The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zuidgeest MGP, Heath M, Lagerwaard B, van Weelij DR, Rutgrink L, Hanke S, Vedenkannas T, Kosonen T, Collamati S, Fons-Martinez J, Veen D, Gardarsdottir H, Mackenzie IS, Dupont S, Grobbee DE; Trials@Home consortium. Bringing Trial Activities to Participants-The Trials@Home RADIAL Proof-of-Concept Trial Investigating Decentralization of Trials. Clin Pharmacol Ther. 2025 Nov;118(5):1037-1045. doi: 10.1002/cpt.70025. Epub 2025 Sep 1. PMID 40888335
- See also: Website Trials@Home project — http://trialsathome.com